CLINICAL TRIAL: NCT05058222
Title: Effect of Deep Breathing Exercises on Post Operative Sleep Duration and Quality in Patients Undergoing CABG (Coronary Artery Bypass Graft).
Brief Title: Effect of Deep Breathing Exercises on Post Operative Sleep Duration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00875 Amna Iqbal
Record Dates: First submitted 2021-03-06; First posted 2021-09-27 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Coronary Artery Bypass Graft
Keywords: Breathing exercises; Coronary artery bypass; Sleep

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep breathing ex (10 reps) Group (Active Comparator): The control program will consist of Deep Breathing Exercises (from Morning to night every three hours; each session consisting of 10 deep breaths with a few seconds pause between each set, for 3 days) in addition with progressive Exercises.
  Interventions: Other: Deep Breathing Exercise after every 3hrs, each session consists of 10 deep breaths Exercise
- Deep breathing ex (30 reps) Group (Experimental): The intervention group will perform additional Deep breathing Exercises (from Morning to night every three hours; each session consisting of 30 deep breaths with a few seconds pause between each set, for 3 days).
  Interventions: Other: Deep Breathing Exercise after every 3hrs, each session consist of 30 deep breaths Exercise

INTERVENTIONS:
Other: Deep Breathing Exercise after every 3hrs, each session consists of 10 deep breaths Exercise — • The control program will consist of Deep Breathing Exercises (from Morning to night every three hours; each session consisting of 10 deep breaths with a few seconds pause between each set, for 3 days) in addition with progressive Exercises.
  Arms: Deep breathing ex (10 reps) Group
Other: Deep Breathing Exercise after every 3hrs, each session consist of 30 deep breaths Exercise — • The intervention group will perform additional Deep breathing Exercises (from Morning to night every three hours; each session consisting of 30 deep breaths with a few seconds pause between each set, for 3 days).
  Arms: Deep breathing ex (30 reps) Group

SUMMARY:
This study will provide the evidence that during the postoperative period deep breathing exercise combined with physical training can positively influence the sleep duration and quality. This study will provide the evidence that during the postoperative period deep breathing exercise combined with physical training can positively influence the sleep duration and quality.

DETAILED DESCRIPTION:
Subjects will be randomly placed into Control group and Interventional group. The control program will consist of Deep Breathing Exercises (from Morning to night every three hours; each session consisting of 10 deep breaths with a few seconds pause between each set, for 3 days) in addition with progressive Exercises. Two daily sessions with an average duration of 25 min will be performed. In addition to the physiotherapeutic program standardized by the hospital's team of physical therapists, the intervention group will perform additional Deep breathing Exercises (from Morning to night every three hours; each session consisting of 30 deep breaths with a few seconds pause between each set, for 3 days). Deep breathing exercises will start 48 hours after extubation and full education along with the routine care (i.e.: from the fourth to sixth postoperative day).

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and write
* Stabilization of vital signs [blood pressure, pulse, respiration)
* Patient undergoing OFF Pump Coronary Artery Bypass Graft (CABG) Procedure

Exclusion Criteria:

* History of severe mental diseases resulting in hospitalization and drug treatment within the previous 6 months
* Use any kind of other complementary methods such as massage therapy, aromatherapy, etc. to treat sleep disorders for the previous two weeks
* History of sleep or respiration disorders and used CNS medications in the night.

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
St Mary's Hospital Sleep Questionnaire (SMHSQ) | Baseline
  To check the quality of sleep over the past 24 hours. This SMH tool was a 14 item multiple choice and short answer instrument which examined individuals' previous nights sleep.
St Mary's Hospital Sleep Questionnaire (SMHSQ) | 3 week
  To check the quality of sleep over the past 24 hours. This SMH tool was a 14 item multiple choice and short answer instrument which examined individuals' previous nights sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Anam Aftab, Phd*, Principal Investigator — Riphah college of rehabilitation and allied health sciences - Rawalpindi
Locations (1):
- Armed forces Institute of Cardiology, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No